CLINICAL TRIAL: NCT06054295
Title: Somatic Mosaicism in Twins Discordant for Childhood Cancer: a Pilot Study
Brief Title: Somatic Mosaicism in Twins Discordant for Childhood Cancer
Status: Recruiting | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AEPI22N2
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Central Nervous System Tumor; Central Nervous System Tumor; Discordant Twin; Somatic Mutation
MeSH Terms: conditions — Central Nervous System Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-Correlative: Twins with CNS tumors, identified through the Children's Oncology Group's Project:EveryChild (PEC) registry, will have both blood and saliva samples collected at the time of study enrollment.
  Interventions: Other: Biospecimen collection; Other: Questionnaire Administration

INTERVENTIONS:
Other: Biospecimen collection — Collection of both blood and saliva samples from participants at the time of study enrollment
Other: Questionnaire Administration — The brief questionnaire will assess health history, demographics, environmental exposures, family history of cancer, and birth characteristics.

SUMMARY:
Somatic mosaicism in cancer associated genes is one potential explanation for discordance in childhood cancer that has not been fully explored to date. This pilot study will focus on twins with central nervous system (CNS) tumors who are identified through the Children's Oncology Group's Project: EveryChild (PEC) registry or volunteer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To conduct a descriptive study of same sex twins (MZ and DZ) discordant for childhood CNS tumors identified through the Children's Oncology Group Project:EveryChild registry.

II. To compare the prevalence of somatic mosaicism in classic cancer-associated genes in monozygotic (MZ) twins discordant for childhood brain tumors. In our pilot study, we will sequence blood and saliva DNA samples from 25 MZ twin pairs using a panel of 94 known cancer associated genes.

SECONDARY OBJECTIVES:

I. To compare the profile of mutations detected in DNA extracted from pre- and post-treatment blood samples from a subset of CNS tumor patients. The purpose of this aim is to ensure that differences in somatic mosaicism detected in twin pairs are not caused by cancer therapy.

Outline:

Twins with CNS tumors will undergo blood and saliva DNA samples with the goal is to learn more about genetic differences that may lead to CNS tumor development.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patient with CNS tumor or have recurrent disease and enrolled on APEC14B1.
* Patient must have same sex twin. Note: (history of) treatment on a COG therapeutic trial is not required.
* Patients must be diagnosed at < 19 years of age at the time of diagnosis.
* A family is eligible to participate if the twin with the CNS tumor is deceased but has a blood sample banked through APEC14B1.
* All patients and/or their parents or legal guardians must provide informed consent. Assent will be obtained for participants between the ages of 8-17 years.
* All institutional, FDA, and NCI requirements for human studies must be met.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Newly diagnosed same sex twins with pediatric central nervous system (CNS) tumors
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Compare the prevalence of somatic mosaicism in classic cancer-associated genes in monozygotic (MZ) twins discordant for childhood brain tumors. | Up to 18 months
  Sequence blood and saliva DNA samples from 25 MZ twin pairs using a panel of 94 known cancer associated genes.

SECONDARY OUTCOMES:
Compare the profile of mutations detected in DNA extracted from pre- and post-treatment blood samples from a subset of CNS tumor patients. | Up to 18 months
  Determine the frequency of somatic mosaicism in twins discordant for CNS tumors. Will use an exact test of proportions to determine whether the affected twin is more likely to have a mosaic mutation. The comparison of pre-treatment and post-treatment samples in the CNS tumor cases will include a descriptive comparison of the mutations identified in each sample

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Poynter, PhD, Study Chair — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States